CLINICAL TRIAL: NCT04492839
Title: The Effect of an Intestinal Adsorbent on Hydrogen and Methane Breath Testing, in Patients With Abdominal and Reflux Symptoms, on Long Term Proton Pump Inhibitor Therapy
Brief Title: Intestinal Adsorbent and Breath Gas Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Anthony Hobson (Other)
Responsible Party: Sponsor-Investigator, Dr Anthony Hobson, Clinical Director, The Functional Gut Clinic
Organization: The Functional Gut Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FGC-19-001
Record Dates: First submitted 2020-07-09; First posted 2020-07-30 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Gastroesophageal Reflux; Small Intestinal Bacterial Overgrowth
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Masking Description: Participants will be masked to the name of the product, but will be informed it is an intestinal adsorbent, class IIa medical device, available to buy over the counter.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intestial adsorbent arm (Experimental): This is a single arm study, all participants will receive the class IIa intestinal adsorbent medical device
  Interventions: Device: Intestinal adsorbent

INTERVENTIONS:
Device: Intestinal adsorbent — Participants will consume the 15ml of the intestinal adsorbent (3.5 g Silicon dioxide in 100 ml Silicic acid gel, Preservatives: Sorbic acid (E 200), Sodium benzoate (E 211). ) three times daily for 10 days. There are no known side effects of the medical device. The product is a class IIa medical device under the European council directive and the product will be used within it's current indications.

SUMMARY:
To determine the effect of an intestinal adsorbent on hydrogen and methane breath levels in patients who have been on long term PPI therapy reporting reflux and abdominal symptoms at baseline.

DETAILED DESCRIPTION:
Participants will be recruited either through clinics at the functional gut clinic or through interest shown to advertising for the study. If the patient is deemed eligible they will be given atleast 24 hours to review the patient information sheet. If they would like to proceed with participation they will be given the chance to ask the study team any questions. If they would still like to proceed the participant will be asked to sign three copies of the informed consent form.

The participants will be required to visit the clinic twice during the study. The day before visit 1 the patient will be required to follow a low residue diet as part of preparation for the hydrogen methane breath. On the day of the first visit participants will complete a hydrogen methane breath test as per the functional gut clinics test protocol, the patient will also be asked to fill two questionnaires about their symptoms. Participants will then be provided with a 10 day bowel and symptom diary and a 10 day supply of blinded the intestinal adsorbent . Participants will be provided with instructions on how to take the the study product and training on completing their daily diary. They will be required to take the study product for 10 consecutive days according to manufacturers instructions.

Participants will return for the second and final visit on the final day of consuming the study product. The day before visit 2 the patient will be required to follow a low residue diet as part of preparation for the hydrogen methane breath. On the day of the second visit participants will complete a hydrogen methane breath test as per the functional gut clinics test protocol, the patient will also be asked to fill two questionnaires about their symptoms. Once these study procedures are complete the participants will have finished their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Participant has provided written informed consent before participating in the study after being given a full description of the study and prior to any study-specific procedures being performed.

  2. Patient has been taking PPI therapy for >6 months 3. Patient reports bloating ≥3 on screening questionnaire 4. Patient reports one of the following ≥3 on screening questionnaire - belching, heartburn, nausea, reflux sensation 5. Participant is a male or non-pregnant female and is age 18 years of age or above 6. Participant is able to communicate well with the Investigator and to comply with the requirements for the entire study.

  7. Participant has capacity to understand written English 8. Participant agrees to follow pre-test diet for 24 hours before giving test sample (Appendix A).

  9. Participant agrees to refrain from strenuous physical activity on the day of the breath test.

  10. Participant agrees to refrain from smoking on the day of the breath test 11. Participant agrees to an overnight fast on the night before the breath test. Food and drink must be withheld until after all breath test samples have been taken.

  12. Participant agrees to not take any probiotic for 7 days before the breath test.

  13. Participant has a body mass index (BMI) between 18.5 and 34.9kg/m2 (bounds included).

Exclusion Criteria:

1. Participant reports using any prohibited medication, medical device or supplementation
2. Participant has taken antibiotics or undergone colonoscopy/sigmoidoscopy in the 4 weeks prior to enrolment.
3. Participant has a diagnosis of any organic gastrointestinal disease, including inflammatory bowel disease, coeliac disease and diverticulitis.
4. Participant has known mechanical obstruction of the GI tract
5. Participant has diabetes
6. Participant has any hepatic disease
7. Participant has any disease of the CNS
8. Participant is involved in this study as an Investigator, sub-Investigator, study coordinator, other study staff, or Sponsor member.
9. Participant has had previous abdominal or colorectal surgery except appendectomy, cholecystectomy, or hysterectomy.
10. Participant has previously taken Silicolgel in the past month
11. Participant has a known hypersensitivity to any of the ingredients of Silicolgel
12. Participant suffers regularly from constipation
13. Participant is involved in any other research projects either currently or during the previous month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
To determine the effect of Silicolgel on hydrogen and methane breath levels in patients who have been on long term PPI therapy reporting reflux and abdominal symptoms at baseline. | 18 months
  Hydrogen and methane breath testing will be used to take readings of participants breath gas levels (hydrogen and methane) as a measure of microbial fermentation.
  Mean change in cumulative total breath hydrogen and methane, will be determined from baseline HMBT to end of study HMBT. Cumulative total hydrogen and cumulative total methane will be calculated independently of one each other. Breath hydrogen and breath methane will be measured in units of parts per million (ppm). Statistical significance will be determined using a paired t-test (p<0.05).
  Each HMBT samples will be analysed using gas chromatography analysis on the day of the breath test being carried out. Breath carbon dioxide will also be measured in order to verify the validity of each sample and apply a correction factor. A correction factor above 2.5 (CO2 < 2%) is considered an invalid sample.

SECONDARY OUTCOMES:
To determine the effect of Silicolgel on abdominal symptoms in patients who have been on long term PPI therapy reporting reflux and abdominal symptoms at baseline. | 18 months
  The IBS-SSS is a validated questionnaire that will be used to determine severity of abdominal and bowel symptoms. The questionnaire is comprised of 7 questions, 5 of which are scored from 0 to 10. The total of these 5 questions will be calculated and multiplied by 10 to determine symptom severity. Mean difference in scores from baseline IBS-SSS and end of study IBS-SSS will be determined using a paired t-test, to determine significance (p<0.05).
To determine the effect of Silicolgel on reflux symptoms in patients who have been on long term PPI therapy reporting reflux and abdominal symptoms at baseline. | 18 months
  The Reflux Questionnaire is a validated questionnaire that will be used to determine severity of upper GI symptoms. The questionnaire is made up of 16 questions, each scored 0 to 5. The total of these 16 questions will be calculated to determine symptom severity. Mean difference in scores from baseline reflux questionnaire and end of study reflux questionnaire will be determined using a paired t-test, to determine significance (p<0.05).

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Hobson, PhD, Principal Investigator — Clinical Director
Locations (1):
- The Functional Gut Clinic, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT04492839/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT04492839/ICF_001.pdf